CLINICAL TRIAL: NCT01689311
Title: In Vitro Myometrial Contractions in Laboring and Non-laboring Women: Oxytocin is Superior to Other Uterotonic Agents
Brief Title: In Vitro Myometrial Contractions in Laboring and Non-laboring Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: University of Toronto (Other); Canadian Anesthesiologists' Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-06; 09-0053-E (Other: REB (MSH))
Record Dates: First submitted 2012-09-17; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Postpartum Hemorrhage
Keywords: Uterine contraction; Dose response; Non-laboring; Laboring; Laboring with oxytocin augmentation; Oxytocin; Ergonovine; Prostaglandin F2alpha; Misoprostol
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — Oxytocin; Ergonovine; Dinoprost; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): All samples will undergo dose response treatment (increasing concentrations) of one of the four uterotonic drugs: oxytocin, ergonovine, prostaglandin F2alpha, or misoprostol.
  Interventions: Drug: Oxytocin; Drug: Ergonovine; Drug: Prostaglandin F2alpha; Drug: Misoprostol

INTERVENTIONS:
Drug: Oxytocin — Oxytocin, 10-10mol/L to 10-5mol/L; solution made in double-distilled autoclaved water and then tested in physiological salt solution.
  Other Names: Pitocin
Drug: Ergonovine — Ergonovine, 10-10mol/L to 10-5mol/L; solution made in double-distilled autoclaved water and then tested in physiological salt solution.
  Other Names: Ergot; Ergometrine
Drug: Prostaglandin F2alpha — Prostaglandin F2alpha, 10-10mol/L to 10-5mol/L; solution made in double-distilled autoclaved water and then tested in physiological salt solution.
Drug: Misoprostol — Misoprostol, 10-10mol/L to 10-5mol/L; solution made in double-distilled autoclaved water and then tested in physiological salt solution.
  Other Names: Synthetic prostaglandin E1

SUMMARY:
The purpose of this study is to compare the ability of an isolated sample of uterine muscle tissue (in a tissue bath) to contract in the presence of various drugs. The drugs studied--uterotonics--are typically used to contract the uterus when a pregnant patient continues to bleed after delivery. Amongst common uterotonic drugs, namely oxytocin, ergonovine, prostaglandin F2alpha, and misoprostol, the most effective one to use is unknown.

The investigators will be testing isolated uterine muscle samples to increasing concentrations of these four drugs in three patient populations: non-laboring, laboring without exogenous oxytocin augmentation, and laboring with oxytocin augmentation. Contractile measures will be measured and compared between all groups. The investigators hypothesize that oxytocin alone will have a weaker uterotonic effect in oxytocin-augmented laboring patients, and all four drugs will induce different patterns of contractions.

DETAILED DESCRIPTION:
Postpartum hemorrhage (PPH) is a major cause of maternal mortality and morbidity. In 80% cases of PPH, the primary cause is failure of the uterus to contract after delivery of the baby, which then requires further treatment of the mother with uterotonic drugs (drugs used to contract uterus and thus prevent bleeding).

Patients participating in this study will be asked to donate a very small sample of uterine tissue during Cesarean section, which will be tested in the laboratory for the ability to contract in response to the uterotonics oxytocin, ergonovine, prostaglandin F2alpha, and misoprostol. We will seek to better understand the effects of these drugs by comparing their contractile capability in isolated uterine tissue.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 37-41 weeks
* Patients requiring primary or first repeat Cesarean section
* Cesarean section under spinal anesthesia

Exclusion Criteria:

* Patients who require general anesthesia
* Patient who had previous myometrial surgery or more than one previous Cesarean section
* Patients with placental anomalies
* Patients with multiple pregnancy (twins, etc.)

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2009-03; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Amplitude of contraction | 4-5 hours

SECONDARY OUTCOMES:
Integrated area under response curve (AUC) | 4-5 hours
Basal tone | 4-5 hours
Frequency of contraction | 4-5 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Balki M, Erik-Soussi M, Kingdom J, Carvalho JC. Comparative efficacy of uterotonic agents: in vitro contractions in isolated myometrial strips of labouring and non-labouring women. Can J Anaesth. 2014 Sep;61(9):808-18. doi: 10.1007/s12630-014-0190-1. Epub 2014 Jun 7. PMID 24906304